CLINICAL TRIAL: NCT00925327
Title: Safety and Effectiveness of the UV-X System for Corneal Collagen Cross-Linking for Compassionate Treatment in Pediatric Patients With Progressive Keratoconus
Acronym: CXL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peschke Meditrade, GmbH (Industry)
Responsible Party: Rudi Peschke, Peschke Meditrade GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVX-004
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Progressive Keratoconus
MeSH Terms: interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Corneal collagen cross-linking with riboflavin and UVA light (Experimental)
  Interventions: Other: Corneal collagen cross-linking with riboflavin/UVA light

INTERVENTIONS:
Other: Corneal collagen cross-linking with riboflavin/UVA light — Corneal collagen cross-linking with riboflavin/UVA light

SUMMARY:
This is a compassionate treatment protocol for the use of the UV-X system for corneal collagen cross-linking (CXL) in eyes with progressive keratoconus in patients who have conditions that limit their capacity to comply with the cross-linking treatment procedures required by ongoing clinical trials.

DETAILED DESCRIPTION:
This is a non-randomized study. All eyes that qualify for the study will receive the cross-linking (CXL) procedure. Corneal collagen cross-linking is performed as a single treatment. Depending on the patient's condition, the CXL procedure may be performed under sedation or anesthesia. Subjects are followed for 12 months after the procedure to evaluate the long term effects of corneal collagen cross-linking.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to 18 years
* Having a diagnosis of progressive keratoconus
* Signed written informed consent
* Having a condition that limits the patient's capacity to comply with the cross-linking treatment procedures and/or the diagnostic tests and measurements required by the ongoing clinical studies
* Willingness and ability to comply with schedule for follow-up visits

Exclusion Criteria:

* Corneal pachymetry at the screening exam that is <400 microns at the thinnest point
* Previous ocular condition in the eye(s) to be treated that may predispose the eye for future complications, for example (herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, or corneal dystrophy, etc.)
* A history of delayed epithelial healing in the eye(s) to be treated
* Pregnancy or lactation during the course of the study
* A known sensitivity to study medications

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Estimated)

PRIMARY OUTCOMES:
Change in keratometry | 3 Months

SECONDARY OUTCOMES:
Change in manifest refraction spherical equivalent | 3 Month

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospitals and Clinics, Kansas City, Missouri, United States